CLINICAL TRIAL: NCT03953170
Title: Pilot Study to Investigate the Effect of Teduglutide on Temporary Ileostomy Function and Complications
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding ended
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, James McCormick, DO, Principal Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Teduglutide
Record Dates: First submitted 2019-04-15; First posted 2019-05-16 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Ileostomy - Stoma
MeSH Terms: interventions — teduglutide; ALX-0600

STUDY DESIGN:
Intervention Model Description: Study subjects will be randomized to Teduglutide or placebo arm in a 1:1 allocation.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The drug will be delivered to the patient according to the randomization scheme and neither the patient nor the investigators will know which patient is randomized into which group until the study is completed. Only the pharmacist at the AHN pharmacy will know the patient assigned to each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Teduglutide (Active Comparator): Teduglutide 0.05 g/kg/day
  Interventions: Drug: Teduglutide
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teduglutide — Teduglutide (Gattex, Shire) was approved by the FDA in 2012 for use in adult patients with short bowel syndrome requiring parenteral support only.
  The results of this study will not be used to justify a change of indication, or dose currently approved for Teduglutide, and will not be used to advertise the drug. This study meets all of the requirements for exemption from the IND regulations and an IND exemption has been confirmed by the FDA.
  Other Names: Gattex
  Arms: Teduglutide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to investigate the natural history of patients with a temporary ileostomy and to assess the effect of Teduglutide in reducing morbidity, hospital readmissions and post reversal complications.

DETAILED DESCRIPTION:
This is a prospective, controlled, randomized, double blind study. A total of 36 subjects will be enrolled into the study. Subjects will be randomized to receive Teduglutide or Placebo for 12 weeks or until the ileostomy is reversed. Teduglutide or placebo will be administered via a daily subcutaneous injection into the abdomen or thigh. The sites will be rotated with each injection. If adverse effects develop the subjects will be permitted to hold drug administration for a maximum of 5 days in total during the 12-week study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing temporary ileostomy (loop or end ileostomy) regardless of the indication or technique used (open or laparoscopy) as part of their regular standard of care
* Age- 18-80 years old
* Normal routine laboratories (CMP, CBC, CRP, amylase, lipase)
* Permitted medications will include biologicals which dose has not been changed for > 6 months, and immunosuppressant therapy which dose has not been changed for 3 months (i.e. codeine sulfate, loperamide, or Lomotil)

Exclusion Criteria:

* Emergency need for ileostomy
* Pregnant or nursing
* Malnutrition or requiring parenteral or enteral nutrition
* Known intestinal obstruction, stricture, or adhesions that would predispose the patient to the development of intestinal obstruction, perforation, hemorrhage, or intestinal abscess
* Intestinal fistulas or abscess proximal to the ostomy
* Small bowel resection greater than 50 cm.
* Clinically significant cardiovascular, renal, pulmonary, endocrine, immunologic, dermatology, neurological or psychiatric disorders
* Cholelithiasis or pancreatitis
* Family history of colorectal cancer or familial polyposis
* Cancer in the last 5 years
* History of HIV, Hepatitis B or C, or other acute systemic or intestinal infections requiring antibiotics
* Use of GLP1 analogues which may increase the risk of acute pancreatitis
* Treatment of Octreotide

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
Change in daily 24 hr ileostomy collection | Change from time of surgery to 12 weeks
  (mL/day)

CONTACTS AND LOCATIONS:
Overall Officials: James McCormick, DO, Principal Investigator — Allegheny Health Network
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
De-identified study data will be shared with study sponsor (Shire Human Genetics Therapies, Inc)